CLINICAL TRIAL: NCT00213161
Title: Establishing an Iron Supplementation Strategy to Reduce the Prevalence of Iron Deficiency Anemia Among Infants and Young Children in India.
Brief Title: Using Iron Supplementation to Decrease Iron Deficiency Anemia in Infants and Young Children in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000001031; CIHR: GLH-63082
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Anemia
Keywords: anemia; iron deficiency; iron drops; iron supplement; malnutrition; pediatrics
MeSH Terms: conditions — Anemia; Iron Deficiencies; Malnutrition | interventions — Iron-Dextran Complex

INTERVENTIONS:
Drug: iron supplement, iron drops

SUMMARY:
The purpose of this study is to determine the smallest dose of Sprinkles, a single-serving package of iron and other micronutrients, to treat infants with iron deficiency anemia in India. Results have implications for programs using Sprinkles worldwide because lower doses of iron may have fewer side effects.

DETAILED DESCRIPTION:
Iron deficiency anemia affects two thirds of children in most developing nations, and even mild anemia can have serious implications for child development. In India, government programs within India have been ineffective in controlling this public health problem due to the lack of effective iron supplements reaching children.

Our research group developed 'Sprinkles', an inexpensive micronutrient supplement which is a single-serve sachet of tasteless powder that contain encapsulated iron and other micronutrients. Parents can be easily instructed to mix the contents of one sachet into a bowl of any complementary food.

This study is part of a partnership and capacity development between interdisciplinary research groups at The Hospital for Sick Children, University of Toronto, Canada and the King Edward Memorial Hospital in India, aimed at developing a long-term program of research that will address iron deficiency anemia among infants and young children in India. For Sprinkles to be implemented into national programs in India, a comprehensive strategy is needed which includes a single, safe and effective iron dose for the Indian population.

This specific study is to conduct a community-based, randomized clinical trial in India to determine the appropriate dose of supplementation required for the target age group.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 months of age
* anemic (Hb 70-100g/L)
* ingesting weaning food in addition to breast milk
* free from major illness (including symptomatic for malaria) and afebrile
* living within study area for the next two months
* parental consent obtained
* only one child per household in the study

Exclusion Criteria:

* Hb < 70 or ≥ 100 g/L
* Not receiving any complementary foods
* Receiving an iron supplement within two weeks of the date of enrolment
* chronic illness
* severely malnourished: weight for age z-score < -3.0
* another child in the household is a subject in this study

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 425
Dates: Start 2004-08; Study Completion 2005-06

PRIMARY OUTCOMES:
Hemoglobin at 4 weeks, 8 weeks, 8 months after first dosing

SECONDARY OUTCOMES:
Ferritin at 8 weeks
Serum Transferrin Receptor (sTfR) at 8 weeks
side effects every 2 weeks
compliance with iron supplement assessed every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Zlotkin, PhD, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- King Edward Memorial Hospital (KEM), Pune, Maharashtra, India